CLINICAL TRIAL: NCT01725347
Title: Validation of a Digital Diet Method for Use With Preschoolers
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor of Pediatric Nutrition, Baylor College of Medicine
Other Study IDs: H-29112; R01CA142919-01A1 (NIH)
Record Dates: First submitted 2012-10-31; First posted 2012-11-12 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Feeding Behaviors
Keywords: nutrition assessment; children; preschool; eating behavior; Head Start; digital technology
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples are to be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- African American Girls: -25% of sample is African American Girls
- African American Boys: -25% of sample is African American Boys
- Hispanic American Girls: -25% of sample is Hispanic American Girls
- Hispanic American Boys: -25% of sample is Hispanic American Boys

SUMMARY:
The Validation of a Digital Diet Method project is very innovative because it links three methods to address the gap in measuring food intake of HS preschool children. Data collection is based on EMA theory; participant burden is low, and the Food Image App decreases participant and staff burden even further. Data management and analysis are semi-automated and relies on advanced computer algorithms. A strength of this approach is its semi-automation, which allows us to leverage the strengths of human operators and computer automation.

DETAILED DESCRIPTION:
The goal of the proposed research is to modify the Remote Food Photography Method (RFPM) for use with preschoolers. Primary caregivers (the majority will be mothers) and HS assistants will use a Smartphone to capture 24-hour images of HS children's food selection and plate waste. The RFPM, Ecological Momentary Assessment (EMA). and the Food Photography Application© will be used to estimate the energy and nutrient intake of preschoolers. The accuracy of the RFPM will be examined by determining the energy and nutrient intake (collectively referred to as food intake [FI]) to established methods: 1) actual gram (g) weights of laboratory-based test meals and 2) doubly labeled water (DLW) in a natural environment.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years old
* Attends Head Start
* African-American
* Hispanic American
* Can physically complete the tasks required in the proposed research

Exclusion Criteria:

* Younger than 3 years old
* Older than 5 years old
* Does not attend Head Start
* Race/Ethnicity other than African-American or Hispanic-American
* Cannot physically complete the tasks required in the proposed research

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: With an anticipated attrition rate of 15%, 62 children will be recruited, resulting in a sample size of 54 after attrition (14 HA boys; 14 HA girls; 13 AA boys; 13 AA girls).
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
This experiment will compare energy intake (EI) calculated using the test method (Remote Food Photography Method or RFPM) against energy intake calculated using weight measures (actual weighing of all food/beverages consumed). | 12 months
  The Bland-Altman method was used to measure the agreement between digital photography estimated weight and actual weight. This method uses a two step process that evaluates the accuracy (validity) of a "new" measurement technique compared to and existing "gold standard", which was the actual weights of foods.

SECONDARY OUTCOMES:
This experiment will compare energy intake (EI) calculated using the test method (Remote Food Photography Method or RFPM) against energy expenditure using the Doubly Labeled Water method (DLW). | 12 months
  The Same statistical analysis methods used for the Primary Outcome Measure will be applied. Additionally, the Bland-Altman technique will be used to assess the degree of agreement between the two methods.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Nicklas, DrPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- USDA/ARS Children's Nutrition Research Center, Houston, Texas, United States

REFERENCES:
- [Result] Nicklas TA, O'Neil CE, Stuff J, Goodell LS, Liu Y, Martin CK. Validity and feasibility of a digital diet estimation method for use with preschool children: a pilot study. J Nutr Educ Behav. 2012 Nov-Dec;44(6):618-23. doi: 10.1016/j.jneb.2011.12.001. Epub 2012 Jun 23. PMID 22727939
- [Derived] Nicklas T, Saab R, Islam NG, Wong W, Butte N, Schulin R, Liu Y, Apolzan JW, Myers CA, Martin CK. Validity of the Remote Food Photography Method Against Doubly Labeled Water Among Minority Preschoolers. Obesity (Silver Spring). 2017 Sep;25(9):1633-1638. doi: 10.1002/oby.21931. Epub 2017 Jul 31. PMID 28758370
- [Derived] Nicklas T, Islam NG, Saab R, Schulin R, Liu Y, Butte NF, Apolzan JW, Myers CA, Martin CK. Validity of a Digital Diet Estimation Method for Use with Preschool Children. J Acad Nutr Diet. 2018 Feb;118(2):252-260. doi: 10.1016/j.jand.2017.05.005. Epub 2017 Jun 19. PMID 28637631